CLINICAL TRIAL: NCT00414817
Title: Phone Calls to Promote Adherence With Inhaled Corticosteroids
Brief Title: Telephone-Based Program to Promote Inhaled Corticosteroid Adherence Among Individuals With Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 443; R01HL083433 (NIH); R01HL083433-01A1 (NIH)
Record Dates: First submitted 2006-12-20; First posted 2006-12-22 (Estimated); Results first posted 2017-01-30 (Estimated); Last update posted 2017-01-30 (Estimated); Status verified 2016-12

CONDITIONS: Asthma
Keywords: Inhaled Corticosteroids; ICS; Adherence
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Automated Phone-Based Refill Reminders (Experimental): Intervention Arm: Participants randomly assigned to this study arm may receive up to 8 automated phone calls from the BREATH EASY Medication Reminder Program over the course of the 19 month intervention period.
  Interventions: Behavioral: Automated Phone-Based Refill Reminders
- Usual Care (No Intervention): Usual Care: Participants randomly assigned to this arm received the same introductory letter as those in the intervention arm, giving them the opportunity to opt out, but were subsequently selected to be in the "usual care" study arm, and therefore, receive no intervention.

INTERVENTIONS:
Behavioral: Automated Phone-Based Refill Reminders — The BREATHE EASY Medication Reminder Program uses interactive voice recognition phone technology to offer timely reminders to patients to refill their ICS medication, educational messages about ICS, and may offer to transfer them to a refill line or to speak with a pharmacist if they have questions.
  Other Names: The BREATHE EASY Medication Reminder Program
  Arms: Automated Phone-Based Refill Reminders

SUMMARY:
Inhaled corticosteroids (ICS) are often prescribed as a treatment for asthma. However, many individuals who take these medications do not adhere to their prescribed treatment regimen. The purpose of this study is to evaluate the effectiveness of a telephone-based program at improving medication adherence among individuals with asthma.

DETAILED DESCRIPTION:
Asthma is a serious, chronic disease that affects lung function and impairs an individual's ability to breathe normally. ICS reduce airway inflammation and are often prescribed to treat these conditions. However, poor medication adherence is a common problem that can lead to treatment failure, hospitalization, or death. A telephone-based system that uses interactive voice recognition technology to remind individuals to follow their medication regimen may prove beneficial in promoting adherence. The purpose of this study is to evaluate the effectiveness of such a telephone-based intervention at improving adherence to inhaled corticosteroid regimens among individuals with asthma. If this study proves successful, telephone-based interventions may be developed to promote treatment adherence for other chronic medical conditions.

This 19-month study will enroll approximately 14,000 members of the Kaiser Permanente Northwest or Hawaii health system. Participants will be randomly assigned to either take part in the telephone intervention or receive usual medical care. Over the 19-month period, participants in the intervention group will receive between one and eight phone calls that will remind them to refill their prescriptions and offer education about ICS. If needed, the call may also offer a transfer to a pharmacy refill line or to speak with a pharmacist. Approximately 2,000 participants will complete questionnaires at study entry and at the end of the 19-month intervention period. The questionnaires will assess quality of life, respiratory health, asthma control, depression, inhaler use beliefs, and satisfaction with the intervention. Electronic medical record data and questionnaires will be used to determine adherence rates.

ELIGIBILITY:
Inclusion Criteria:

* Received treatment for asthma in the year prior to study entry
* Received at least one respiratory medication at a Kaiser Permanente Northwest (KPNW) or Kaiser Permanente Hawaii (KPH) outpatient pharmacy in the year prior to study entry
* Continuous Kaiser Permanente membership from the year prior to study entry through study entry
* Willing to participate in the study

Exclusion Criteria:

* Excluded from primary analyses if fewer than three months of follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14064 (Actual)
Dates: Start 2007-06; Primary Completion 2009-04 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William M. Vollmer, PhD, Principal Investigator — Center for Health Research/KPNW; Cynthia Rand, PhD, Principal Investigator — Johns Hopkins University; Joan Dubanoski, PhD, Principal Investigator — Center for Health Research/KPH; Adrianne Feldstein, MD, Principal Investigator — Center for Health Research/KPNW; David Smith, PhD, Principal Investigator — Center for Health Research/KPNW
Locations (2):
- United States (2):
  - Center for Health Research/KPH, Honolulu, Hawaii
  - Center for Health Research-KPNW, Portland, Oregon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vollmer WM, Xu M, Feldstein A, Smith D, Waterbury A, Rand C. Comparison of pharmacy-based measures of medication adherence. BMC Health Serv Res. 2012 Jun 12;12:155. doi: 10.1186/1472-6963-12-155. PMID 22691240
- [Result] Vollmer WM, Feldstein A, Smith DH, Dubanoski JP, Waterbury A, Schneider JL, Clark SA, Rand C. Use of health information technology to improve medication adherence. Am J Manag Care. 2011 Dec;17(12 Spec No.):SP79-87. PMID 22216772
- [Result] Schneider J, Waterbury A, Feldstein A, Donovan J, Vollmer WM, Dubanoski J, Clark S, Rand C. Maximizing acceptability and usefulness of an automated telephone intervention: Lessons from a developmental mixed-methods approach. Health Informatics J. 2011 Mar;17(1):72-88. doi: 10.1177/1460458210391220. PMID 25133772
- See also: main outcomes, Amer J Manag Care 2011 — http://www.ncbi.nlm.nih.gov/pubmed/22216772
- See also: Vollmer et al, BMC Hlth Serv Res 2012. contains further details on computation of primary outcome measure and its performance characteristics — http://www.ncbi.nlm.nih.gov/pubmed/22691240

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred, starting in October 2007 via electronic medical record query. Calling campaigns ended in April 2009.
Pre-assignment Details: 14,064 adults taking medication for asthma were pre-randomized to intervention or usual care (UC). However, only those individuals who ever qualified for an intervention call were included in the analysis sample. This included 6905 pre-existing inhaled corticosteroid (ICS) users (our primary analysis sample) and 1612 new ICS users.
Groups:
- Automated Phone-Based Refill Reminders: Intervention Arm: Participants randomly assigned to this study arm may receive up to 8 automated phone calls from the BREATH EASY Medication Reminder Program over the course of the 19 month intervention period.
  Automated Phone-Based Refill Reminders : The BREATHE EASY Medication Reminder Program uses interactive voice recognition phone technology to offer timely reminders to patients to refill their ICS medication, educational messages about ICS, and may offer to transfer them to a refill line or to speak with a pharmacist if they have questions.
Period: Overall Study
Arm/Group | Automated Phone-Based Refill Reminders | Usual Care
Started | 7033 | 7031
Never Started on ICS | 1465 (Not initial users of ICS and not starting during study, hence don't qualify for analysis sample.) | 1392 (Not initial users of ICS and not starting during study, hence don't qualify for analysis sample.)
Died or Left Health Plan | 451 (These individuals died or terminated Health Plan membership prior to ever qualifying for a call.) | 417 (These individuals died or terminated Health Plan membership prior to ever qualifying for a call.)
Adherent ICS User | 922 (Fully adherent ICS users who never qualified for an intervention call.) | 900 (Fully adherent ICS users who never qualified for an intervention call.)
Daily Oral Steroid User | 117 (qualified for analysis sample, but excluded due to subsequent determination of oral steroid use.) | 123 (qualified for analysis sample, but excluded due to subsequent determination of oral steroid use.)
<3 Months Follow-up | 175 (qualified for analysis sample, but excluded since follow-up too short to assess adherence reliably.) | 184 (qualified for analysis sample, but excluded since follow-up too short to assess adherence reliably.)
Completed | 3903 (Qualified for primary analysis (3171 prior ICS users) or secondary analysis (732 new users) samples.) | 4015 (Qualified for primary analysis (3260 prior ICS users) or secondary analysis (755 new users) samples.)
Not Completed | 3130 | 3016

BASELINE CHARACTERISTICS:
Population: individuals who met our inclusion/exclusion criteria
Groups:
- Automated Phone-Based Refill Reminders: Intervention arm participants who were included in the primary outcome analysis. This consists of existing users of inhaled corticosteroids at the outset of the study, qualified (or for UC would have qualified) for an intervention call at some point during the study, had at least 3 months of follow-up, and were not subsequently determined to be daily oral steroid users.
- Usual Care: usual care participants who were included in the primary outcome analysis. This consists of existing users of inhaled corticosteroids at the outset of the study, qualified (or for UC would have qualified) for an intervention call at some point during the study, had at least 3 months of follow-up, and were not subsequently determined to be daily oral steroid users.
- Total: Total of all reporting groups
Arm/Group | Automated Phone-Based Refill Reminders | Usual Care | Total
Number analyzed (Participants) | 3171 | 3260 | 6431
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2394 | 2499 | 4893
  >=65 years | 777 | 761 | 1538
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.7 (15.3) | 53.5 (15.3) | 53.6 (15.3)
Gender [Count of Participants; unit: Participants]
  Female | 2150 | 2207 | 4357
  Male | 1021 | 1053 | 2074
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 43 | 39 | 82
  Not Hispanic or Latino | 1169 | 1185 | 2354
  Unknown or Not Reported | 1959 | 2036 | 3995
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 16 | 20 | 36
  Asian | 342 | 388 | 730
  Native Hawaiian or Other Pacific Islander | 145 | 130 | 275
  Black or African American | 51 | 52 | 103
  White | 1632 | 1578 | 3210
  More than one race | 196 | 235 | 431
  Unknown or Not Reported | 789 | 857 | 1646
Region of Enrollment [Number; unit: participants]
  United States | 3171 | 3260 | 6431

OUTCOME MEASURES:

1. Primary Outcome: Modified Medication Possession Ratio
Description: We used a modification of the Medication Possession Ratio (MPR) as our primary outcome measure. The MPR is computed as the number of days' supply of medication dispensed during a given time window divided by the time between the first dispensing in the window and the end of the window. Our modified MPR (mMPR) also accounted for medication that was on hand at the start of the window and ignored any days' supply that would extend beyond the end of the window. The MPR, and by extension the mMPR, assumes that medications were used as directed and that a new inhaled corticosteroid canister was not started until any medication on hand was exhausted.
Time Frame: Measured over 19 months
Population: Study participants who were existing users of ICS at the outset of the study, qualified (or for UC would have qualified) for an intervention call at some point during the study, had at least 3 months of follow-up, and were not subsequently determined to be daily oral steroid users.
Measure: Mean (Standard Deviation); unit: fraction of days with medication
Arm/Group | Automated Phone-Based Refill Reminders | Usual Care
Number analyzed (Participants) | 3171 | 3260
fraction of days with medication | .40 (.32) | .38 (.32)
Statistical Analysis 1: Comparison: Automated Phone-Based Refill Reminders vs Usual Care; In all of our analyses we used duration of follow-up as a weighting variable to reflect the fact that our adherence measure becomes more accurate and reliable with longer follow-up. This weighting is reflected both in the formal statistical analyses and in the presentation of means and standard deviations given above. Also, sensitivity analyses that included daily oral steroid users and those with fewer than 3 months of follow-up yielded similar results to those presented here; Test type: Superiority or Other; p = .002, Regression, Linear; 2-tailed p-value based on linear regression adjusted for site, age, sex, co-morbid COPD, baseline use of short acting beta agonists, and baseline mMPR; Mean Difference (Final Values) = 0.018, 95% CI 2-sided [.006 to .030] — Estimated adherence was approximately 2 percentage points higher for intervention group than for usual care group

2. Secondary Outcome: Juniper Asthma Quality of Life Questionnaire (Global Score)
Description: Asthma specific quality of life measurement developed by Dr. Elizabeth Juniper. This is the overall summary score and ranges from 1=poorest quality of life to 7=best quality of life.
Time Frame: Measured at 19 months
Population: We assessed this outcome on a random sample of study participants that over-sampled intervention participants. All were existing users of ICS at the outset of the study who qualified for an intervention call at some point during the study, had at least 3 months of follow-up, and were not subsequently determined to be daily oral steroid users.
Measure: Mean (Standard Deviation); unit: unitless scale ranging from 1-7
Arm/Group | Automated Phone-Based Refill Reminders | Usual Care
Number analyzed (Participants) | 921 | 501
unitless scale ranging from 1-7 | 4.8 (1.3) | 4.9 (1.3)
Statistical Analysis 1: Comparison: Automated Phone-Based Refill Reminders vs Usual Care; In all of our analyses we used duration of follow-up as a weighting variable. This weighting is reflected both in the formal statistical analyses and in the presentation of means and standard deviations given above; Test type: Superiority or Other; p = 0.175, Regression, Linear; 2-tailed p-value adjusted for site, age, sex, co-morbid COPD, baseline use of short acting beta agonists, and baseline adherence; Mean Difference (Final Values) = -0.10, 95% CI 2-sided [-0.23 to 0.04]

3. Secondary Outcome: Rate of Acute Health Care Visits for Asthma
Description: annualized rate of acute asthma health care utilization events (urgent care, emergency department use, hospitalization) based on data derived from the electronic medical record. Each type of event was given equal weight for this analysis.
Time Frame: Measured over 19 months of follow-up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: number of events per year
Arm/Group | Automated Phone-Based Refill Reminders | Usual Care
Number analyzed (Participants) | 3171 | 3260
number of events per year | 1.7 (2.3) | 1.7 (2.0)
Statistical Analysis 1: Comparison: Automated Phone-Based Refill Reminders vs Usual Care; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.852, overdispersed Poisson regression — 2-tailed p-value based on overdispersed Poisson regression adjusted for site, age, sex, co-morbid COPD, baseline use of short acting beta agonists, and baseline mMPR; Risk Ratio (RR) = 1.00, 95% CI 2-sided [0.96 to 1.06]

ADVERSE EVENTS:
Arm/Group | Automated Phone-Based Refill Reminders | Usual Care
Serious Adverse Events (participants affected / at risk) | 0/7033 | 0/7031
Other Adverse Events (participants affected / at risk) | 0/7033 | 0/7031

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No